CLINICAL TRIAL: NCT06157021
Title: Evaluation of Obturation Quality in Necrotic Primary Molars After Manual Versus Rotary Pulpectomy; a Randomized Clinical Trial
Brief Title: Obturation Quality in Primary Molars
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rasha Adel Ragab, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-11-23
Record Dates: First submitted 2023-11-12; First posted 2023-12-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Necrotic Primary Molars
Keywords: Rotary instrumentation; pulpectomy; primary molars; obturation quality

STUDY DESIGN:
Intervention Model Description: Randomized controlled parallel double blinded study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding to the child participants and legal guardian of each participating child, inter examiner and statistician. The operator and the child were blinded to the intervention from the beginning till finishing the procedure of caries removal and access cavity. Blinding cannot be done during root canal instrumentation because of visual differences between manual and rotary files.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotary pulpectomy (Experimental): Rotary pulpectomy using rotary files (Fanta AF baby* rotary files and Endo Radar* rotary device
  Interventions: Procedure: Rotary pulpectomy
- Manual pulpectomy (Active Comparator): Manual pulpectomy using manual H files, Mani*)
  Interventions: Procedure: Manual pulpectomy

INTERVENTIONS:
Procedure: Rotary pulpectomy — Pulpectomy procedures by making cleaning and shaping of root canals of necrotic primary molars using (Fanta AF baby* rotary files and Endo Radar* rotary device).
  Other Names: (Fanta AF baby* rotary files and Endo Radar* rotary device).
  Arms: Rotary pulpectomy
Procedure: Manual pulpectomy — Pulpectomy procedures by making cleaning and shaping of root canals of necrotic primary molars using Manual H files, Mani*)
  Other Names: Manual H files, Mani*)
  Arms: Manual pulpectomy

SUMMARY:
Forty cases of necrotic primary molars in children aged 4-8 years were selected to compare the effect of manual versus rotary pulpectomy regarding parental acceptance and obturation quality.

DETAILED DESCRIPTION:
The present study was performed in the Department of Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University, Egypt.

Ethical approval was obtained from the Ethical Committee board of Faculty of Dentistry, Cairo University, Egypt.

Written informed consent was taken from the legal guardian of each participating child willing to participate in the trial, prior to the start of the clinical procedure after explaining the whole procedure in a simple way. The consent form was written in Arabic.

A sample of 40 primary mandibular second molars of children between 4 and 8 years of age indicated for pulpectomy participated in this double-blinded randomized controlled trial. Parallel allocation design was adopted for the intervention and control arms with allocation ration 1: 1 (i.e. 20 cases each). The sample size was calculated considering the previously published studies with 95% power in detecting the true statistical significance among the two groups.

Control group one: Manual pulpectomy using) H files, Mani*) Group two: Rotary pulpectomy using (Fanta baby* rotary files and Endo Radar* rotary device).

Diagnosis:

Diagnostic chart was filled with personal, medical and dental history.

1. Intra & extra oral examination was made with aid of mirror and probe to assess the clinical inclusion criteria.
2. Preoperative photographs were taken
3. Preoperative radiograph were examined

Intervention:

Patients were assigned into two groups; Group A (Experimental group) (using rotary files)

1. Pre-operative radiograph showing all roots and their apices.
2. Local anaesthetic (to enable use of rubber dam clamp).
3. Rubber dam isolation.
4. Removal of caries.
5. Removal of roof of pulp chamber.
6. Identify root canals.
7. Irrigate with concentrated sodium hypochlorite followed by normal saline (0.9%)
8. Estimate working lengths of root canals keeping 2 mm short of the radiographic apex.
9. Insert rotary files into canals and debride the canals lightly and gently.
10. Irrigate the root canals.
11. Dry canals with pre-measured paper points, keeping 2 mm from root apices.
12. Canals were dried with paper points, obturated by injecting Metapex. (Meta Biomed - Metapex Root Canal Filling Material)
13. Stainless steel crown was performed

Group B (control group) (using manual files) All steps as that of group A were done except step (j) instead of it; a manual files were inserted into the canals for debridement lightly and gently.

Randomization &Allocation concealment:- Sequence generation Simple randomization was done by computer software (www.random.com) for patient's assignment in each group.

Blinding:

Blinding to the child participants and legal guardian of each participating child, inter examiner and statistician.

Statistical analysis:

Categorical data were presented as frequencies (n) and percentages (%). Intergroup comparisons were done utilizing Fisher's exact test. while intragroup comparisons were done utilizing Cochran's Q tests followed by Dunn's post hoc test. Ordinal data were presented as median and interquartile range values and were analyzed using Mann-Whitney U test for intergroup comparisons. The significance level was set at p ≤ 0.05 for all tests. Statistical analysis was performed with ® SPSS® (SPSS Inc., IBM Corporation, New York, USA) Statistics Version 26 for Windows.

ELIGIBILITY:
Inclusion Criteria:

* Medically free children.
* Age: 4-8 years
* Primary molars with necrotic pulp, abscess or fistula.
* Teeth which if lost possibility of space maintainer construction exists.
* Pre-operative radiograph showing absence of root resorption more than one third of the root.

Exclusion Criteria:

* Vital primary teeth.
* Teeth with inadequate tooth structure to support the rubber dam.
* Expected shedding time within one year.
* Peri-radicular involvement extending to the permanent tooth bud.
* Excessive internal& external root resorption,
* Perforation of pulpal floor.
* Extensive tooth mobility

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
parental acceptance | Immediately after the intervention
  done by the participating parents who ranked their acceptance to pulpectomy procedures on a five-point Likert scale, as follows: 1, strongly acceptable; 2, acceptable; 3, neutral; 4, unacceptable; and 5, strongly unacceptable. (Scores from 1-3 means better outcome)

SECONDARY OUTCOMES:
obturation quality | Immediately after the intervention and after 6 months
  (Postoperative radiograph was used to determine obturation quality as (secondary outcome) using Coll and Sadrian criteria (Coll and Sadrian, 1996) at baseline postoperatively and after 6 months.
  Coll and Sadrian criteria define the root canal obturation quality as optimal fill, underfill, or overfill. Underfill means that all the canals were filled 1 mm or more short of the apex, optimal fill means that one or more canals have filling material ending at radiographic apex, and overfill means any canal showing filling material outside the root. Optimum filled means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Rasha A Ragab, Lecturer, Principal Investigator — Faculty of Dentistry, Cairo University, Egypt.
Locations (1):
- Faculty of Dentistry, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
No plan to share